CLINICAL TRIAL: NCT06888323
Title: Lintuzumab-Ac225 Monotherapy for Patients With Hypomethylating Agent-Refractory Myelodysplastic Syndrome
Brief Title: Testing an Anti-cancer Radio-Active Immunotherapy Called Lintuzumab Ac225 in Patients With High-Risk Myelodysplastic Syndrome That Has Not Responded to Other Treatment
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug Supply Issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-01929; NCI-2025-01929 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10695 (Other: Dana-Farber - Harvard Cancer Center LAO); 10695 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Actinium; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lintuzumab-ac225) (Experimental): Patients receive lintuzumab-ac225 IV, over 30 minutes, on day 1 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo SPECT/CT scans and buccal swab on study, as well as bone marrow aspiration throughout the trial.
  Interventions: Radiation: Actinium Ac 225 Lintuzumab; Procedure: Bone Marrow Aspiration; Procedure: Buccal Swab; Procedure: Computed Tomography; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Radiation: Actinium Ac 225 Lintuzumab — Given IV
  Other Names: 225Ac-HuM195; Actimab-A; Actinium (225Ac) Lintuzumab Satetraxetan; Actinium-225-Labeled Humanized Anti-CD33 Monoclonal Antibody HuM195; LINTUZUMAB SATETRAXETAN AC-225; SGN-33 AC-225
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Buccal Swab — Undergo buccal swab
  Other Names: Buccal Scraping; Buccal Smear; Buccal swab/scraping; Buccal Swabbing
Procedure: Computed Tomography — Undergo SPECT/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase I trial tests the safety, side effects and best dose of lintuzumab-ac225 for the treatment of patients with high risk myelodysplastic syndrome that has not responded to previous treatment (refractory). Lintuzumab-ac225 is a monoclonal antibody, called lintuzumab, linked to a radioactive agent called Ac225. Lintuzumab attaches to CD33 positive cancer cells in a targeted way and delivers Ac225 to kill them. Giving lintuzumab-ac225 may be safe, tolerable and/or effective in treating patients with high risk, refractory myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, tolerability, and maximum tolerated dose of actinium ac 225 lintuzumab (lintuzumab-ac225) monotherapy in myelodysplastic syndrome/neoplasm (MDS) patients whose disease is refractory to or progressing on hypomethylating agent (HMA) therapy.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the efficacy, complete remission (CR) (CR/complete remission with incomplete bone marrow recovery [CRi]) rates, overall response rates (ORR), progression free survival (PFS), and overall survival (OS) of lintuzumab-Ac225 in MDS patients whose disease is refractory to or progressing on HMA therapy.

III. To perform bulk ribonucleic acid (RNA) sequencing to assess transcriptomic changes in MDS patients after HMA therapy.

IV. Dosimetry studies V. To study the correlation of absorbed radiation doses (in Gy) with adverse events and disease control.

OUTLINE: This is a dose-escalation study of lintuzumab-ac225 followed by a dose-expansion study.

Patients receive lintuzumab-ac225 intravenously (IV), over 30 minutes, on day 1 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo single photon emission computed tomography (SPECT)/CT scans and buccal swab on study, as well as bone marrow aspiration throughout the trial.

After completion of study treatment, patients are followed for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of MDS by bone marrow biopsy by World Health Organization (2016) guidelines
* Patients with MDS who have progressed or had no response after 6 cycles of azacitidine or 4 cycles of decitabine

  * For the expansion phase, we will be enrolling 12 more patients at the maximum tolerated dose: 6 patients with prior azacitidine or decitabine treatment and 6 patients with prior treatment with azacitidine or decitabine in combination with venetoclax
* Patients with MDS must have ≥ 5% myeloblasts
* Patients with demonstration of CD33 positive myeloblasts on flow cytometry using Phycoerythrin (PE) labeled anti-CD33 antibody, done as standard of care testing by every participating site
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of lintuzumab-Ac225 in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Serum direct bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN
* Creatinine clearance ≥ 50mL/min (Cockcroft-Gault equation)
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* The effects of lintuzumab-Ac225 on the developing human fetus are unknown. For this reason and because CD33 radiotherapy agents are known to be teratogenic, female patients of childbearing age must have had a negative serum pregnancy test within 14 days of initiation of dosing and must agree to use of two acceptable methods of birth control while on the study drug. A woman must agree to remain on a highly effective method throughout the study and for at least 6 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. During the study and for 30 days after receiving the last dose of study drug in addition to the highly effective method of contraception, a man (a) who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (e.g. condom with spermicidal foam/gel/film/cream/suppository); (b) who is sexually active with a woman who is pregnant must use a condom; (c) must agree not to donate sperm
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients have active clinically significant graft vs. host disease (GVHD) or are on systemic corticosteroids
* Patients have clinically active central nervous system (CNS) leukemia
* Patients who are receiving any other investigational agents, such as experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is shorter, prior to enrollment, or is currently enrolled in any other type of medical research (e.g. medical device) not scientifically or medically compatible with this study
* Patients who are receiving any therapy that can result in increased toxicity on this study or confound the study findings, within the last 30 days or 5 half-lives, whichever is shorter, prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lintuzumab-Ac225
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make this protocol unreasonably hazardous
* Pregnant women are excluded from this study because lintuzumab-Ac225 is a CD33 radiotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lintuzumab-Ac225, breastfeeding should be discontinued if the mother is treated with lintuzumab-Ac225
* The patient had major surgery within 14 days prior to enrollment
* No prior radiopharmaceutical therapy and no radiation therapy within the last 120 days prior to cycle 1 day 1 (C1D1), as this may contribute to added toxicity
* Patients who are unable to take spironolactone or eplerenone due to intolerance, allergy, drug-drug interactions, or for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-27 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 70 days from first dose of lintuzumab-ac225

SECONDARY OUTCOMES:
Complete remission rate | Up to 90 days after completion of treatment
  Calculated as per the 2023 myelodysplastic syndrome (MDS) response criteria.
Overall response rate | Up to 90 days after completion of treatment
  Calculated as per the 2023 MDS response criteria.
Progression free survival | Up to 90 days after completion of treatment
  Calculated as per the 2023 MDS response criteria.
Overall survival | Up to 90 days after completion of treatment
  Calculated as per the 2023 MDS response criteria.
Transcriptomic changes | At baseline and after cycle 2 (cycles = 28 days)
  Ribonucleic acid sequencing analysis will be performed from cryopreserved bone marrow samples.
Incidence of adverse events | Up to 90 days after completion of treatment
  Will be graded using Common Terminology Criteria for Adverse Events 5.0 and described by frequency, duration, and severity of treatment-emergent, treatment-related, and serious adverse events. All reported toxicities, regardless of attribution, will be summarized by toxicity type and maximum grade, and sorted by number of patients experiencing the toxicity for each dosing cohort and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Talha Badar, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (1):
- Dana-Farber - Harvard Cancer Center LAO, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm